CLINICAL TRIAL: NCT05967299
Title: A Phase 1 Single-Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Intravenous ZMA001 in Healthy Subjects
Brief Title: Study of Intravenous ZMA001 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Zymedi, Co., Ltd. (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 10001522; 001522-H
Record Dates: First submitted 2023-07-27; First posted 2023-08-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12-05

CONDITIONS: Pulmonary Arterial Hypertension PAH
Keywords: human monoclonal antibody (IgG1)
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Cohort 1 (1.5 mg/kg/dose) only (Placebo Comparator): Placebo for ZMA001 is supplied in a single-use 10 mL glass vial. Each vial contains 30 mg/mL of sucrose.Placebo drug is manufactured using the same ingredients as active drug (20 mM histidine-HCl buffer [pH 5.6], 30 mg/mL sucrose, 0.070 w/v% polysorbate 80) excluding ZMA001 antibody and is packed in the same vial.
  Interventions: Other: Placebo Cohort 1 (1.5 mg/kg/dose) only
- ZMA001 (BC-NKA-20008) (Experimental): ZMA001 is a fully human, monoclonal antibody (IgG1) that inhibits migration of activated monocytes and macrophages and reduces pulmonary vascular remodeling and pulmonary artery pressure in pre-clinical rodent models of pulmonary arterial hypertension (PAH).
  Interventions: Drug: ZMA001 (BC-NKA-20008)

INTERVENTIONS:
Other: Placebo Cohort 1 (1.5 mg/kg/dose) only — 30mg/ml Sucrose
  Arms: Placebo Cohort 1 (1.5 mg/kg/dose) only
Drug: ZMA001 (BC-NKA-20008) — ZMA001 is a fully human, monoclonal antibody (IgG1) that inhibits migration of activated monocytes and macrophages and reduces pulmonary vascular remodeling and pulmonary artery pressure in pre-clinical rodent models of pulmonary arterial hypertension (PAH).
  Arms: ZMA001 (BC-NKA-20008)

SUMMARY:
Background:

A number of diseases can cause a type of lung injury called pulmonary arterial hypertension (PAH). Most people who develop PAH do not survive more than a few years. A new study drug (ZMA001) may help. ZMA001 is a monoclonal antibody. This type of drug consists of proteins, made in a facility, that are very similar to proteins in a human body. But before giving ZMA001 to people sick with PAH, researchers want to find out how the drug affects healthy people.

Objective:

To test a drug (ZMA001) in healthy volunteers.

Eligibility:

Healthy adults aged 18 to 60 years.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have a urine test for drug use. They will have a test of their heart function.

Participants will come to the clinic for 1 inpatient visit of up to 48 hours.

ZMA001 is a liquid administered through a tube attached to a needle inserted into a vein in the arm. Participants will receive this drug only once, during their inpatient stay. Some participants will receive the drug; others will receive a placebo in Cohort 1 only. A placebo is a treatment that looks just like the real drug but contains no medicine. Participants will not know which treatment they are getting in Cohort 1. Cohorts 2-4 will receive a single dose of the study drug, administered through a tube attached to a needle inserted into a vein in the arm.

After a screening visit, participants will have 1 inpatient visit and up to 8 outpatient visits over 16 weeks after receiving the treatment. Blood draws and other tests will be repeated. Each outpatient visit is approximately 2 hours long.

This study is the first time ZMA001 will be administered to people.

DETAILED DESCRIPTION:
Study Description:

ZMA001 is a fully human, monoclonal antibody (IgG1) that inhibits migration of activated monocytes and macrophages and reduces pulmonary vascular remodeling and pulmonary artery pressure in pre-clinical rodent models of pulmonary arterial hypertension (PAH). The current first-in-human, single ascending-dose study will determine the safety, tolerability, and pharmacokinetics of intravenous ZMA001 in healthy subjects.

Objectives:

Primary Objective: Safety and tolerability of ZMA001 in healthy subjects

Secondary Objectives: Determine the pharmacokinetics of ZMA001 in healthy subjects following a single, intravenous dose

Endpoints:

Primary Endpoint: The number of all-cause, treatment-emergent adverse events, grade 1 and above (following CTCAE v5.0 criteria) through day 113

Secondary Endpoints: For each ZMA001 dose level (1.5, 0.25, 0.50, and 1.0 mg/kg), the following will be determined [Timeframe: Pre-infusion, end of infusion, 2, 4, 8, 12, 24, and 48h; Days 8, 15, 22, 29, 57, 85 and 113]:

1. Time to peak drug concentration (Tmax)
2. Peak drug concentration (Cmax)
3. Area under the drug concentration-time curve (AUC)
4. Elimination half-life

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male* or female, aged 18 to 60 years, inclusive
3. In good general health as evidenced by medical history
4. Females of childbearing potential agree to use an accepted method of contraception (see below) throughout study participation and for 120 days after study drug infusion.
5. Males sexually active with a female partner must agree to use a condom with spermicide for 120 days after study drug infusion or be surgically sterile for at least 90 days before screening. Males must also agree to not donate sperm for 120 days after study drug administration.
6. Agreement to adhere to Lifestyle Considerations throughout study duration
7. Ability of subject to understand and the willingness to sign a written informed consent document.

   * Enrollment of healthy male subjects will be limited to no more than 14 out of the total study cohort of 32 in order to ensure an adequate representation of female subjects.

Accepted methods of contraception for females of childbearing potential:

* Use of an implanted or intrauterine hormonal device for at least 30 consecutive days before study drug infusion
* Use of oral, patch or injectable contraceptives or a vaginal hormonal device for at least 30 consecutive days before study drug infusion
* Use of a non-hormonal intrauterine device for at least 30 consecutive days before study drug infusion
* Two barrier methods such as a diaphragm with spermicide or a condom with spermicide

EXCLUSION CRITERIA:

An individual who meets any of the following criteria prior to informed consent will be excluded from participation in this study:

1. Pregnancy or lactation. Females of childbearing potential must have a negative serum Beta-human chorionic gonadotropin test no more than 48 hours from study drug infusion.
2. A history of human immunodeficiency virus (HIV) infection.
3. History of severe drug or excipient allergy or hypersensitivity
4. Known allergy to any of the components of the investigational drug or placebo
5. Recent infection or febrile illness within the past 14 days
6. Treatment with another investigational drug within the past 30 days or 5 half-lives, whichever is longer
7. Any vaccination within the past 4 weeks or receipt of a live-attenuated vaccine within the past 6 months
8. Use of tobacco products within the past 3 months
9. Illicit drug use (e.g. cocaine, opioids, methamphetamine, PCP) within the past 6 months or positive urine drug screen at Screening Visit
10. Marijuana (cannabis) use within the past 30 days or positive urine drug screen at Screening Visit
11. History of alcohol abuse within the past 2 years
12. Current clinically significant medical illness that is uncontrolled despite appropriate medical treatment including (but not limited to) hematologic, oncologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, infectious, hepatic, dermatologic, psychiatric, neurologic, autoimmune or allergic disease
13. Body mass index less than 17 or greater than 32 kg/m^2
14. Clinically significant abnormal results on clinical blood testing completed at the Screening Visit
15. Electrocardiographic evidence of clinically relevant heart disease
16. Diabetes mellitus requiring medical treatment
17. Received another monoclonal antibody in the past 30 days
18. Use of herbal supplements, or similar products within the past 2 weeks
19. Blood donation equal to or above 500 mL within 2 months prior to dosing.
20. Any other finding that, in the judgment of the Investigator, would increase the risk of having an adverse outcome from participating in the study.

Justification to exclude minors: Given that the vast majority of patients with PAH are >18 years of age and the fact that this is a first in human study, the risks of including children/minors (ie. subjects < 18 yrs of age) are not justified given the limited potential benefits of including these subjects.

Justification to exclude adults >60 years old: Subjects > 60 years of age are more likely to have comorbid medical conditions that could place them at increased risk of participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of ZMA001 in healthy subjects | day 113
  The number of all-cause, treatment-emergent adverse events, grade 1 and above (following CTCAE v5.0 criteria) through day 113

SECONDARY OUTCOMES:
Determine the pharmacokinetics of ZMA001 in healthy subjects following a single, intravenous dose. | Pre-infusion, end of infusion, 2, 4, 8, 12, 24, and 48h; Days 8, 15, 22, 29, 57, 85 and 113
  For each ZMA001 dose level (1.5, 0.25, 0.50, and 1.0 mg/kg), the following will be determined.3. Area under the drug concentration-time curve(AUC)
Determine the pharmacokinetics of ZMA001 in healthy subjects following a single, intravenous dose. | Pre-infusion, end of infusion, 2, 4, 8, 12, 24, and 48h; Days 8, 15, 22, 29, 57, 85 and 113
  For each ZMA001 dose level (1.5, 0.25, 0.50, and 1.0 mg/kg), the following will be determined.2. Peak drug concentration (Cmax)
Determine the pharmacokinetics of ZMA001 in healthy subjects following a single, intravenous dose. | Pre-infusion, end of infusion, 2, 4, 8, 12, 24, and 48h; Days 8, 15, 22, 29, 57, 85 and 113
  For each ZMA001 dose level (1.5, 0.25, 0.50, and 1.0 mg/kg), the following will be determined.1. Time to peak drug concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Elinoff, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of associated publication and the duration of availability is expected to be indefinite but will ultimately be determined by the NHLBI.@@@@@@
Access Criteria: Data will be shared through the NHLBI BioData Catalyst, which is a controlled access repository.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001522-H.html